CLINICAL TRIAL: NCT05112978
Title: Evaluation of Patellar Dimension and Bristol Index in Asian Population: an MRI Study
Brief Title: Evaluation of Patellar Dimension and Bristol Index in Asian Population
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ismail Hadisoebroto Dilogo, Prof, Indonesia University
Other Study IDs: BRIS
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Patello Femoral Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — MRI genu non contrast

SUMMARY:
Restoration of patellar thickness is pivotal during a total knee arthroplasty (TKA). Several studies showed there are differences in the knee measurements between Asian and Western population. This study aims to evaluate the patellar dimension and Bristol Index of patellar width to thickness (BIPWiT) using magnetic resonance imaging (MRI) in Asian population.

ELIGIBILITY:
Inclusion Criteria:

* knee pain

Exclusion Criteria:

* degenerative joint disease
* patellofemoral pathology

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: all patients came to clinic
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
bristol index | 1 day MRI examination

SECONDARY OUTCOMES:
patellar sizes | 1 day MRI examination

CONTACTS AND LOCATIONS:
Locations (1):
- Pondok Indah Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No